CLINICAL TRIAL: NCT03991845
Title: A Randomised Controlled Trial to Evaluate the Effect of Vitamin D Supplementation in Patients With Chronic Urticaria
Brief Title: A Trial to Evaluate the Effect of Vitamin D Supplementation in Patients With Chronic Urticaria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Davinder Parsad, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INT/IEC/2017/1314
Record Dates: First submitted 2018-01-29; First posted 2019-06-19 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Urticaria; Vitamin D Deficiency
MeSH Terms: conditions — Urticaria; Vitamin D Deficiency | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose Vit D (Experimental): All Patients belonging to arm 1 will be treated with low dose oral Vit D (2000 IU/day) for 12 weeks
  Interventions: Drug: Vit D
- High dose Vit D (Active Comparator): All patients in this group will be treated with high dose oral Vit D (60,000 IU/week) for 12 weeks
  Interventions: Drug: Vit D
- Placebo (No Intervention): No Vit D supplementation will be given to patients in this group

INTERVENTIONS:
Drug: Vit D — Vit D supplementation was done
  Other Names: Levocetirizine 10 mg once daily will be given to all patients
  Arms: High dose Vit D; Low dose Vit D

SUMMARY:
This study will be an assessor-blind, randomized controlled trial in patients with CSU. The investigators will compared Vit D level in patients with Chronic spontaneous urticaria (CSU) and controls. Enrolled CSU patients with Vit D level <30ng/ml will be then randomized into three intervention arms in the ratio of 1:1:1. Patients belonging to intervention group A will be treated with low dose Vit D (2000 IU/day) for 12 weeks according to the Indian council of medical research (ICMR) guidelines. Intervention group B patients will be treated with high dose Vit D (60,000 IU/week) for 12 weeks and group C will not be given any Vit D supplements. All patients will be evaluated after 12 weeks. The urticaria activity score over 4 days (UAS4) will be used to assess the disease severity using the number of wheals and pruritus intensity based on the EAACI/GA2LEN/EDF guidelines. The patient's disease severity levels will be graded as mild (0-8), moderate (9-16), and severe (17-24).

DETAILED DESCRIPTION:
This is a prospective, randomized, single-centre clinical study. Serum Vit D level will be assessed in all patients at baseline. Patients with Vit D level ≥30 will be excluded from the trial but included in the study and those with Vit D level <30 will be randomized into 3 groups A, B and C. Patients with Vit D level ≥30 will be categorized into Group D. Patients belonging to Group A will be treated with low dose Vit D (2000 IU/day) according to Indian council of medical research (ICMR) guidelines. Those in Group B will be treated with high dose Vit D (60,000 IU/week) and group C will not be given any Vit D supplements. Patients belonging to Group A and B will be treated for 12 weeks in order to safely restore Vit D and achieve a steady state. In addition levocetirizine, 10 mg will be given to all patients in groups to control urticaria symptoms. All patients will be treated according to EAACI/GA2LEN/EDF guidelines after 12 weeks. All participants will also be provided with rescue prednisone use for intolerable or uncontrolled symptoms. At 6 weeks and 12 weeks, a physician assessment (physician blinded to treatment arm) will be conducted to check if patients had intolerable symptoms or took rescue prednisolone 40 mg therapy. Safety monitoring will be completed throughout the entirety of the study. Specific stopping rules and discontinuation of the study included pregnancy, a serum Vit D level higher than 100 ng/mL, or a serum calcium level higher than 11 mg/dL. Patients will be followed for 6 weeks after the study completion and thereafter data analysis will be done in 3 steps:

Step 1: Comparison of serum Vit D level in CSU patients vs. controls Step 2 : Assessment of factors associated with Vit D deficiency in urticaria patients Step 3: Effect of Vit D supplementation (group A (low dose), group B (high dose), group C(no supplementation) on urticaria severity using UAS4

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age, having urticaria episodes at least 2 days per week for 6 weeks or longer with/without angioedema.

Exclusion Criteria:

* Patients with only physical urticaria, only dermatographism, urticarial vasculitis, hereditary or acquired angioedema.
* Patients with BMI>25 kg/m2, dyslipidemia, diabetes, hypertension, pre-existing cardiovascular disease, cerebro-vascular accidents, hypothyroidism, smokers, and other systemic or cutaneous disorders including atopic dermatitis, psoriasis etc.
* Patients with hypercalcemia (>11 mg/dL), diabetes, renal insufficiency, hepatic disorders, hyperparathyroidism, sarcoidosis, other granulomatous disorders, malignancy.
* Pregnant and lactating women, patients who have taken Vit D supplementation in past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2019-11-27 (Estimated); Study Completion 2019-12-28 (Estimated)

PRIMARY OUTCOMES:
Change in Urticaria Activity Score- UAS 4 | upto 12 weeks
  Urticaria activity score (UAS) over previous 4 days i.e 4 days before starting treatment and second reading after 12 weeks. It includes calculation of wheals and itching over past 4 days on a scale of 0-3 making a total score of 6 per day and total score of 24 of past 4 days. Maximum score 24, minimum score 0, range 0-24. No subscale will be assessed . 0 indicated no disease and 24 indicates maximum severity. The readings will be taken before and after treatment completion. Change in UAS before starting treatment, and at 12 weeks follow-up visit will be used to assess the efficacy of intervention. Intervention will be stopped at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Davinder Parsad, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-06-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03991845/Prot_ICF_000.pdf